CLINICAL TRIAL: NCT03923881
Title: Multispectral Optoacoustic Imaging Using Cetuximab-800CW for Detection of Cervical Lymph Node Metastases: a Single Center Proof of Concept Study
Brief Title: MSOT Using Cetuximab-800CW for Detection of Cervical Lymph Node Metastases
Acronym: OPUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, dr. M.J.H. Witjes, Principal Investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL67343.042.18
Record Dates: First submitted 2019-04-17; First posted 2019-04-23 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Oral Cancer; Lymph Node Metastases
Keywords: Multispectral Optoacoustic Tomography; Molecular Imaging; Cetuximab-800CW
MeSH Terms: conditions — Mouth Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Intervention Model Description: 20 patients that have been included in the ICON-study (NCT03134846) and therefore will be administered with cetuximab-800CW
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients with oral squamous cell carcinoma that have been included in ICON-study and are scheduled for treatment of neck
  Interventions: Device: MSOT Acuity Echo

INTERVENTIONS:
Device: MSOT Acuity Echo — Optoacoustic imaging with the MSOT Acuity Echo
  Other Names: Administration of cetuximab-800CW as part of the ICON-study (NCT03923881)

SUMMARY:
The presence of lymph node metastasis is an important factor in determining the appropriate treatment plan in patients with OSCC. However, detection of lymph node metastases by means of current imaging modalities is limited. 20-30% of patients with a clinically negative neck (cN0) harbour lymph node metastasis that were not detected during clinical diagnostic workup, which are referred to as occult lymph node metastasis. Therefore, patients with a risk of lymph node metastasis higher than 20% undergo a sentinel node procedure (SNP) or elective neck dissection (END), which means that a substantial part of patients is overtreated. There is need for an additional non-invasive diagnostic tool that can identify lymph node metastasis and thereby support the decision making for treatment of the neck.

The main objective of this study is to evaluate if EGFR-positive cervical lymph node metastasis can be detected non-invasively with multispectral optoacoustic imaging using cetuximab-800CW as contrast agent in patients with oral squamous cell carcinoma.

DETAILED DESCRIPTION:
Background: The presence of lymph node metastasis is an important factor in determining the appropriate treatment plan in patients with OSCC. However, detection of lymph node metastases by means of current imaging modalities is limited. 20-30% of patients with a clinically negative neck (cN0) harbour lymph node metastasis that were not detected during clinical diagnostic workup, which are referred to as occult lymph node metastasis. Personalized management of the neck would benefit greatly from staging techniques that increase the accuracy of the assessment of nodal disease. In addition, visualizing the pattern of lymphatic spread can possibly lead to more targeted neck dissections and thereby reduce morbidity. Clearly, there is need for additional diagnostic tools in order to identify lymph node metastasis and thereby support the decision making for treatment of the neck.

Optoacoustic imaging is a novel imaging method in which an ultrashort laser pulse is used to irradiate biological tissue. Consequently, optoacoustic or photoacoustic waves are generated which can be measured by wideband ultrasonic transducers. Optoacoustic imaging has been shown to address clinically relevant aspects of various cancers by enabling visualization of targeted tumor-specific biomarkers by detecting optoacoustic waves. We hypothesize that accumulation of cetuximab-800CW can be detected in lymph node metastasis, enabling better visualization of regional metastatic disease compared to current imaging modalities. This approach can improve detection of lymph node metastases and thereby supports decision making for treatment of the neck.

Objectives: The main objective of this study is to evaluate if EGFR-positive cervical lymph node metastasis can be detected non-invasively using the MSOT Acuity Echo with cetuximab-800CW as contrast agent in patients with oral squamous cell carcinoma.

Study design: The current study is a single center, prospective, cross-sectional, proof of concept study. The study will be carried out by the out at the University Medical Center Groningen, Department of Oral and Maxillofacial Surgery and Department of Nuclear Medicine and Molecular Imaging. Further analysis of sections of the lymph node metastasis will be done at the Department of Pathology.

Study population: 20 patients with oral squamous cell carcinoma that have been included in the ICON-study (NCT03134846) and are scheduled for treatment of the neck will be included.

Patient related study procedures: Prior to tracer administration as part of the ICON study, optoacoustic imaging is performed. Two-four days later, surgical procedure will take place. One day prior to surgery, the patient is admitted to the hospital and optoacoustic imaging is performed with cetuximab-800CW as contrast agent.

Main study endpoints: Quantification of the cetuximab-800CW optoacoustic signal and tracer distribution observed by multispectral optoacoustic imaging using the MSOT Acuity Echo in vivo in patients with oral squamous cell carcinoma.

Burden, risks and benefit to participation: Time investment: Patients need to visit the UMCG 2-4 days before their planned surgery according to the ICON-study which will take approximately 2 hours. For the first imaging session, the imaging procedure will take 20-30 minutes and therefore the visit is prolonged with 20-30 minutes. Usually patients are admitted one day prior to surgery. Therefore the second imaging on this day will not require extra time investment, although the imaging procedure takes 20-30 minutes Extra procedures: Two imaging procedures, prior to tracer administration and on day of admission. Both imaging procedures will take 20-30 minutes.

Several measures described below have been taken to reduce the risk of injuries to an absolute minimum. The residual risk of MSOT is slight, reversible reddening and temperature increase of the skin.

Patients will have no direct benefit from this study.

ELIGIBILITY:
Inclusion Criteria: patients must meet inclusion criteria of the ICON study (NCT03134846), which are as follows:

* Biopsy confirmed diagnosis of primary or recurrent HNSCC and scheduled to undergo surgical resection as decided by the Multi-Disciplinary Head & Neck Tumor Board of the UMCG.
* Age ≥ 18 years
* Written informed consent
* Adequate potential for follow up
* Acceptable hematologic status, kidney function, and liver function, as standard surgery protocol requires.

Exclusion Criteria:patients must meet exclusion criteria of the ICON study (NCT03134846), which are as follows:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent;
* Concurrent uncontrolled medical conditions;
* Received an investigational drug within 30 days prior to the dose of cetuximab-800CW;
* Tumors at sites of which the surgeon would assess that in vivo imaging would not be feasible;
* Had within 6 months prior to enrollment: myocardial infarction, cerebrovascular accident, uncontrolled cardiac heart failure, significant liver disease, unstable angina;
* Inadequately controlled hypertension with or without current antihypertensive medications;
* History of infusion reactions to cetuximab or other monoclonal antibody therapies
* Pregnant or lactating women. Documentation of a negative pregnancy test must be available for women of childbearing potential. Woman of childbearing potential are premenopausal women with intact reproductive organs and women less than two years after menopause;
* Evidence of QT prolongation on pretreatment ECG (greater than 440 ms in males or greater than 450 ms in females);
* Lab values that in the opinion of the primary surgeon would prevent surgical resection;
* Patients receiving Class IA (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents;
* Magnesium, potassium and calcium deviations that might lead to cardiac rhythm (grade II or higher deviations by CTCAE);
* Life expectancy < 12 weeks;
* Karnofsky performance status < 70%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Optoacoustic signal | A week after imaging is performed
  The optoacoustic signal intensity in lymph nodes compared to surrounding tissue

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No